CLINICAL TRIAL: NCT02821338
Title: A Randomized, 2-Sequence, 2-Treatment, 4-Period, Open-Label, Single Dose, Fully Replicated Comparative Bioavailability Crossover Study of Two Formulations of Lamotrigine Extended Release Tablets in Healthy Subjects Under Fed Conditions
Brief Title: A Bioavailability Crossover Study of Two Formulations of Lamotrigine Extended Release Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Vince & Associates Clinical Research, Inc. (Other); Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15-099D
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: Bioequivalence; Lamotrigine Extended Release; Generic; Pharmacokinetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Active Comparator): The treatments will be administered according to a randomly assigned pre-generated sequence involving the randomized, four-period, two sequence, fully replicate crossover design. Two study drugs involved are: Lamotrigine Extended Release (generic) and Lamictal XR (brand).
  Interventions: Drug: Lamotrigine Extended Release
- Sequence 2 (Active Comparator): The treatments will be administered according to a randomly assigned pre-generated sequence involving the four-period, two sequence, fully replicate crossover design. Two study drugs involved are: Lamotrigine Extended Release (generic) and Lamictal XR (brand).
  Interventions: Drug: Lamotrigine Extended Release

INTERVENTIONS:
Drug: Lamotrigine Extended Release — Lamotrigine Extended Release (generic) and Lamictal XR (brand).
  Other Names: Lamictal XR

SUMMARY:
The objective of this study is to determine bioequivalence between two different formulations of lamotrigine extended release tablets (one reference product and one generic product) in a healthy adult population, following a single oral dose under fed conditions.

DETAILED DESCRIPTION:
This is a single center, randomized, open-label, single dose, two treatment, four-period, two-sequence, fully replicated crossover design in the fed state.

The study will include two treatments:

* Treatment-A: One dose of Lamotrigine extended-release tablet (Test) administered in the morning after a 10-hour overnight fast and 30 minutes after the start of a high-fat, high-calorie breakfast.
* Treatment-B: One dose of Lamictal XR extended-release tablet (Reference) administered in the morning after a 10 hour overnight fast and 30 minutes after the start of a high-fat, high-calorie breakfast.

A total of 30 healthy subjects will be dosed to ensure that at least 24 subjects will complete the 4-period replicate design. For each treatment period, subjects will be confined from the day prior to dosing until approximately 48 hours post-dose. Subjects will return to the clinical site for the remaining blood samples. There will be a minimum 14-day washout between doses.

Subject participation from the Screening Visit to the Follow-Up Visit will be approximately 71 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects ≥18 to ≤50 years of age
2. Subject is willing and able to provide informed consent
3. Body mass index (BMI) greater than or equal to 18.00 kg/m2 and below 30.00 kg/m2 at screening
4. Body weight greater than or equal to 50 kg at screening
5. Subject is a non-smoker and has not used any nicotine containing products within 6 months prior to screening
6. Subjects who are considered generally healthy upon completion of medical history, physical examination, vital signs, screening laboratory results and screening ECG in the opinion of the Investigator
7. Subjects who are willing and able to comply with the visit schedule, laboratory tests, pharmacokinetic sampling schedule and other study procedures
8. Subjects who are willing and able to maintain their eligibility throughout the study.
9. A female study subject must meet one of the following criteria:

   * If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first administration of the study medication, during the study, and for at least 30 days after the last dose of the study medication. An acceptable method of contraception includes one of the following:

     * Abstinence from heterosexual intercourse
     * Progestogen-containing hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
     * Intrauterine device (without hormones)
     * Condom with spermicide
   * If a female of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses), as confirmed by FSH levels (post menopausal must be confirmed by the subject having a serum follicle stimulating hormone greater than 40mIU/ml at screening). Females of non-childbearing potential must present a proof of partial or total hysterectomy; if such proof is not available, the female will be considered to be of childbearing potential.
10. A male study subject must agree to use one of the accepted contraceptive regimens during the study and for at least 90 days after the last dose of the study medication;

    * Abstinence from heterosexual intercourse
    * Female partner with hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
    * Female partner with intrauterine device (with or without hormones)
    * Female partner with condom with spermicide used by male study subject
    * Female partner of non-childbearing potential
    * Male sterilization with absence of sperm in the post vasectomy ejaculate
11. A male study subject must agree not to donate sperm during the study and for at least 90 days after the last dose of the study medication

Exclusion Criteria:

1. Females who are pregnant or are breastfeeding
2. Females who are using any estrogen-containing hormonal contraceptives
3. History of known clinically significant drug allergies or reactions to lamotrigine, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs in the opinion of the Investigator
4. Clinically significant history or evidence of gastrointestinal, hepatic, renal, endocrine, pulmonary, neurological, psychiatric, cardiovascular, hematologic, dermatologic, immunologic disease or any other condition known to interfere with the absorption, distribution, metabolism or distribution of drugs that in the opinion of the Investigator would jeopardize the safety of the subject or impact validity of study results
5. Presence of observed abnormality (evidenced from physical examination, ECG, vital signs, or laboratory evaluation) that would be clinically significant in the opinion of the Investigator
6. History of regular alcohol consumption exceeding 7 drinks per week for females and 14 drinks per week for males within 6 months of screening
7. Has current or recent history (within the past year) of alcohol or drug abuse or dependence
8. Any clinically significant illness in the previous 30 days prior to screening
9. Use of any enzyme-modifying drugs, including strong inhibitors of CYP enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin, St John's Wort) in the previous 30 days prior to screening
10. Known presence of rare hereditary problems of galactose and /or lactose intolerance or glucose-galactose malabsorption
11. Unusual dietary habits (e.g., vegan, Atkins), dietary restrictions, and/or food allergies.
12. Any planned surgery from the screening visit until the end of the study
13. Positive urine screen for alcohol, cotinine and/or drugs of abuse at screening and at each admission of each treatment period
14. Positive test results for HIV-1/HIV-2 Antibodies, Hepatitis B surface Antigen (HBsAg) or Hepatitis C Antibody (HCVAb)
15. Albumin values less than 4 g/dL at screening
16. Triglyceride values greater than 200 mg/dL at screening
17. Treatment with any investigational drug 30 days prior to screening
18. Participation in other clinical studies within 30 days prior to screening
19. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to screening
20. Subject is unlikely to comply with the study protocol or, in the opinion of the Investigator, would not be a suitable candidate for participation in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Vince, D.O., Principal Investigator — Vince and Associates Clinical Research
Locations (1):
- Vince and Associates Clinical Research, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical site — http://www.vinceandassociates.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 (Test-Ref-Test-Ref): Sequence 1 - ABAB. The study was a single center, randomized, open-label, single dose, 2-treatment, 4-period, 2-sequence, fully replicated, crossover design in healthy male and female subjects. All completed subjects received two rounds of Lamictal and Lamotrigine.
  The following investigational products were administered in the fed state:
  Treatment A: A single 1-tablet dose of Lamotrigine 200 mg extended-release tablet (Test) Treatment B: A single 1-tablet dose of Lamictal XR 200 mg extended-release tablet (Reference)
- Sequence 2 (Ref-Test-Ref-Test): Sequence 2 - BABA. The study was a single center, randomized, open-label, single dose, 2-treatment, 4-period, 2-sequence, fully replicated, crossover design in healthy male and female subjects. All completed subjects received two rounds of Lamictal and Lamotrigine.
  The following investigational products were administered in the fed state:
  Treatment A: A single 1-tablet dose of Lamotrigine 200 mg extended-release tablet (Test) Treatment B: A single 1-tablet dose of Lamictal XR 200 mg extended-release tablet (Reference)
Period: Overall Study
Arm/Group | Sequence 1 (Test-Ref-Test-Ref) | Sequence 2 (Ref-Test-Ref-Test)
Started (All completed subjects received two rounds of Lamictal and Lamotrigine.) | 15 | 15
Completed | 12 (12 out of 15 subjects assigned to Sequence 1 completed the study, and provided two data points.) | 13 (13 out of 15 subjects assigned to Sequence 2 completed the study, and provided two data points.)
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: 30 participants
  Completed subjects received two rounds of Lamictal and Lamotrigine.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 32 [20 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.05 (2.54)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Lamotrigine Concentration vs. Time Curve From Sample Time Point 0 Hour to Sample Time Point 144 Hour.
Description: Pre-dose, and post-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36, 48, 72, 96, 120, 144 hours
  Lamotrigine and Lamictal have the same active ingredient "Lamotrigine."
Time Frame: 144 hours
Population: Fully replicated crossover study (all completed subjects received two rounds of Lamictal and Lamotrigine). Completed participants contributed two data points for each treatment, however, some subjects provided one or partial data point.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Units Other Than Participants: data points
Groups:
- Generic Lamotrigine Extended Release Tablet: Lamotrigine Extended Release (generic)
- Brand Lamictal XR Tablet: Lamictal XR (brand)
Arm/Group | Generic Lamotrigine Extended Release Tablet | Brand Lamictal XR Tablet
Number analyzed (Participants) | 24 | 24
Number analyzed (data points) | 44 | 45
h*ng/mL | 119966.6 (32391.0) | 121969.5 (33663.6)
Statistical Analysis 1: Comparison: Generic Lamotrigine Extended Release Tablet vs Brand Lamictal XR Tablet; 90% confidence interval of the geometric mean ratio of test/reference; Test type: Equivalence — 90% confidence interval falls within 80.00-125.00%; Test/Reference ratio = 0.9863, 90% CI 2-sided [0.9598 to 1.0134]

2. Primary Outcome: AUC 0-Inf
Description: Area Under the Lamotrigine Concentrations vs. time curve from sample time point 0 hour to sample time point 144hours plus extrapolation to infinity of the terminal concentration slope. This describes the total exposure to Lamotrigine. Sampling times include: Pre-dose, and post-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36, 48, 72, 96, 120, 144 hours.
  Lamotrigine and Lamictal have the same active ingredient.
Time Frame: 144 hours
Population: Fully replicated crossover design (all completed subjects received two rounds of Lamictal and Lamotrigine). Completed participants contributed two data points for each treatment, however, some subjects provided one or partial data point.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Units Other Than Participants: data points
Arm/Group | Generic Lamotrigine Extended Release Tablet | Brand Lamictal XR Tablet
Number analyzed (Participants) | 24 | 24
Number analyzed (data points) | 43 | 44
h*ng/mL | 128824.9 (39291.6) | 134410.3 (47446.8)
Statistical Analysis 1: Comparison: Generic Lamotrigine Extended Release Tablet vs Brand Lamictal XR Tablet; Test type: Equivalence — 90% confidence interval falls within 80.00-125.00%; Test/Reference Ratio = 0.9785, 90% CI 2-sided [0.9484 to 1.0095]

3. Primary Outcome: Cmax
Description: The maximum concentration of the Lamotrigine achieved in specified time frame for each treatment. Sampling times include: post-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36, 48, 72, 96, 120, 144 hours.
  Lamotrigine and Lamictal have the same active ingredient.
Time Frame: 2 to 144 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: Data points
Arm/Group | Generic Lamotrigine Extended Release Tablet | Brand Lamictal XR Tablet
Number analyzed (Participants) | 24 | 24
Number analyzed (Data points) | 45 | 46
ng/mL | 2338.9 (353.2) | 2244.6 (341.2)
Statistical Analysis 1: Comparison: Generic Lamotrigine Extended Release Tablet vs Brand Lamictal XR Tablet; Test type: Equivalence — 90% confidence interval falls within 80.00-125.00%; Test/Reference Ratio = 1.0470, 90% CI 2-sided [1.0079 to 1.0877]

4. Other Pre Specified Outcome: Tmax
Description: Time from 0 concentration sample point to the Cmax sample point. Sampling times include: post-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36, 48, 72, 96, 120, 144 hours.
Time Frame: 2 to 144 hours
Population: Fully replicate crossover design (all completed subjects received two rounds of Lamictal and Lamotrigine). Completed participants contributed two data points for each treatment, however, some subjects provided one or partial data point.
Measure: Median (Full Range); unit: hours
Units Other Than Participants: data points
Arm/Group | Generic Lamotrigine Extended Release Tablet | Brand Lamictal XR Tablet
Number analyzed (Participants) | 24 | 24
Number analyzed (data points) | 45 | 46
hours | 10 [4 to 27] | 22 [10 to 48]

5. Other Pre Specified Outcome: λZ
Description: Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve. Sampling times include: post-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36, 48, 72, 96, 120, 144 hours.
Time Frame: 2 to 144 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: per hour
Units Other Than Participants: data points
Arm/Group | Generic Lamotrigine Extended Release Tablet | Brand Lamictal XR Tablet
Number analyzed (Participants) | 24 | 24
Number analyzed (data points) | 43 | 44
per hour | 0.0218 (0.0067) | 0.0221 (0.0067)

6. Other Pre Specified Outcome: Thalf
Description: It is the terminal elimination half-life, calculated as ln(2)/λZ. Sampling times include: post-dose 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36, 48, 72, 96, 120, 144 hours.
Time Frame: 2 to 144 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Units Other Than Participants: data points
Arm/Group | Generic Lamotrigine Extended Release Tablet | Brand Lamictal XR Tablet
Number analyzed (Participants) | 24 | 24
Number analyzed (data points) | 43 | 44
hours | 34.77 (10.57) | 34.56 (11.34)

ADVERSE EVENTS:
Arm/Group | Generic Lamotrigine Extended Release Tablet | Brand Lamictal XR Tablet
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 9/30 | 11/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Lamotrigine Extended Release Tablet (N=30) | Brand Lamictal XR Tablet (N=30)
Blood Pressure Systolic Increased (Investigations) | 2 (2) | 1 (1)
Drug Screen Positive (Investigations) | 2 (2) | 1 (1)
Heart Rate Increased (Investigations) | 1 (1) | 1 (1)
Liver Function Test Increased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vessel Puncture Site Pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less